CLINICAL TRIAL: NCT01957215
Title: A Clinical Study to Assess the Efficacy of Pain Relief of Topical Indomethacin Patch Over Placebo in Ankle Sprain Patients
Brief Title: Efficacy of Topical Indomethacin Patch Over Placebo in Ankle Sprain Pain Relief
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Rundo International Pharmaceutical Research & Development Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202177; RH01778 (Other: GSK)
Record Dates: First submitted 2013-10-04; First posted 2013-10-08 (Estimated); Results first posted 2015-06-15 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-04

CONDITIONS: Ankle Sprain
MeSH Terms: conditions — Ankle Injuries | interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Indomethacin patch (Experimental): Indomethacin patch to be applied on the sprained ankle twice a day (BID).
  Interventions: Drug: Indomethacin
- Placebo patch (Placebo Comparator): Placebo patch to be applied on the sprained ankle BID.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Indomethacin — Topical indomethacin
  Arms: Indomethacin patch
Drug: Placebo — Placebo patch
  Arms: Placebo patch

SUMMARY:
This study will investigate the efficacy of the Indomethacin patch in pain relief of ankle sprain in adult patients, compared to a placebo patch

DETAILED DESCRIPTION:
Indomethacin is a non-steroidal anti-inflammatory drug (NSAID) which reduces pain, fever, stiffness and swelling in acute skeletal musculature injuries involving joints. However, oral Indomethacin formulations predisposes for some systemic side effects. To avoid the systemic side effects of oral Indomethacin, a topical Indomethacin formulations have been developed and approved in some countries as an Over the counter product. Present study is to investigate the efficacy of the Indomethacin patch in pain relief of ankle sprain in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Participant with Grade I or Grade II acute sprain of the lateral ankle within 24 hours before screening visit
* Participant with self-assessed pain intensity score after movement (5 steps) at the site of the ankle sprain that is >= 5 as measured on a 0-10 NRS rating.
* Participant with a peri-malleolar edema (sub-malleolar perimeter difference of >=20mm between injured and uninjured ankle)

Exclusion Criteria:

* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Participant who had medication that could interfere with the subject's perception of pain since experiencing ankle sprain.
* Pregnancy , Breast Feeding and Substance Abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- China (15):
  - Changzhou NO.2 People's Hospital, Changzhou, Jiangsu
  - Changzhou NO.2 People?s Hospital, Changzhou, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Ruijin Hospital Luwan Branch, Shanghai, Shanghai Municipality
  - Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai Xuhui Centre Hospital, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Tenth People?s Hospital, Shanghai, Shanghai Municipality
  - Shanghai Tenth Peoples Hospital, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai First People?s Hospital, Shanghai, Shanghai Municipality
  - Shanghai First Peoples Hospital, Shanghai, Shanghai Municipality

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted across multiple sites in China.
Groups:
- Indomethacin Patch: 0.35% w/w Indomethacin patch was applied on the sprained ankle twice a day (BID).
- Placebo Patch: Placebo patch was applied on the sprained ankle BID.
Period: Overall Study
Arm/Group | Indomethacin Patch | Placebo Patch
Started | 135 | 135
Completed | 122 | 123
Not Completed | 13 | 12
Not completed — Adverse Event | 2 | 2
Not completed — Lost to Follow-up | 3 | 3
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Indomethacin Patch: Indomethacin patch was applied on the sprained ankle BID
- Total: Total of all reporting groups
Arm/Group | Indomethacin Patch | Placebo Patch | Total
Number analyzed (Participants) | 135 | 135 | 270
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.7 (12.73) | 35.6 (12.29) | 36.6 (12.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 73 | 149
  Male | 59 | 62 | 121

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Difference (SPID)1-3 Days
Description: SPID was calculated as sum of products of Pain Intensity Differences (PID) at a given time-point (t) with the time-interval from that time-point to the previous time-point (t-1). The time-intervals used were 0 hrs (Day 1, pre treatment), 0.5 hrs, 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, 36 hrs and 48 hrs. Positive and higher scores indicate greater reduction in pain. SPIDt = ∑PID x (time t - time t-1).
  Pain Intensity was assessed at baseline and at each time-point based on numerical rating scale (NRS) which is a horizontal line with a scale from 0-10, where 0 represents "No" and 10 represents the "worst possible pain"
Time Frame: Baseline (Day 1) to Day 3
Population: Efficacy analysis was conducted on the Intent-to-Treat (ITT) population, defined as those participants who received study treatment and had at least one post-baseline efficacy measurement
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Indomethacin Patch | Placebo Patch
Number analyzed (Participants) | 135 | 135
Score on scale | 3.981 (0.2163) | 3.264 (0.2163)
Statistical Analysis 1: Comparison: Indomethacin Patch vs Placebo Patch; Test type: Superiority or Other; p = 0.0201, ANCOVA — P- value was obtained from ANCOVA model with treatment and site as fixed effects and NRS Baseline value as a covariate; Adjusted Mean Difference = 0.72, 95% CI [0.1134 to 1.3199] — ADJ DIFF is the Treatment difference defined as the Adjusted Mean of 0.35% Indomethacin Patches minus Adjusted Mean of Placebo Patches

2. Secondary Outcome: Pain Relief Score (PRS) on Movement Over Time
Description: PRS was assessed for pain on movement (walking 5 steps on flat surface) at 30, 60 minutes and 2, 4, 8 and 12 hrs after the first dose of treatment (indomethacin or placebo patch) and twice daily during the period from 12 hours to 24 hr, 36 hr, 48 hr, 60 hr, 72 hr, 84 hr, 96 hr, 108 hr, 120 hr, 132 hr and 144 hr between treatment groups.
  Participants were asked to choose a number on a scale of 0 to 4, where, 0- No pain relief; 1- A little or perceptible pain relief; 2- Meaningful pain relief; 3- A lot of relief; 4- Complete relief. The mean PRS scores were calculated on the basis of participant's response based on the above score.
Time Frame: 30 minutes (mins) to 144 hours (hrs) post treatment
Population: Efficacy analysis was conducted on ITT population, defined as those participants who received study treatment and had at least one post-baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Indomethacin Patch | Placebo Patch
Number analyzed (Participants) | 135 | 135
Score on scale
  0.5 hours | 0.24 (0.539) | 0.21 (0.546)
  1 hr | 0.40 (0.665) | 0.42 (0.775)
  2 hr | 0.58 (0.806) | 0.53 (0.791)
  4 hr | 0.80 (0.862) | 0.68 (0.942)
  8 hr | 0.84 (0.820) | 0.68 (0.861)
  12 hr | 1.22 (0.900) | 0.94 (1.006)
  24 hr | 1.64 (0.933) | 1.29 (1.055)
  36 hr | 1.93 (0.950) | 1.55 (1.093)
  48 hr | 1.94 (0.963) | 1.63 (1.006)
  60 hr | 2.09 (0.965) | 1.65 (0.988)
  72 hr | 2.18 (0.934) | 1.69 (1.006)
  84 hr | 2.33 (0.886) | 1.84 (0.995)
  96 hr | 2.37 (0.920) | 1.84 (1.018)
  108 hr | 2.36 (0.856) | 2.07 (0.989)
  120 hr | 2.46 (0.954) | 1.97 (1.026)
  132 hr | 2.47 (0.928) | 2.14 (1.072)
  144 hr | 2.56 (0.895) | 2.16 (0.982)

3. Secondary Outcome: NRS for Pain on Movement Over Time
Description: NRS was assessed for pain on movement (walking 5 steps on flat surface) at 30, 60 minutes and 2, 4, 8 and 12 hrs after the first dose of treatment (indomethacin or placebo patch) and twice daily during the period from 12 hours to 24 hr, 36 hr, 48 hr, 60 hr, 72 hr, 84 hr, 96 hr, 108 hr, 120 hr, 132 hr and 144 hr between treatment groups.
  The NRS is a horizontal line with a scale from 0-10. After application of patch (indomethacin or reference patch), patients were asked to choose a number that relates to their pain intensity on the scale of 0 to 10, where 0 represents no pain and 10 represents the worst possible pain.
Time Frame: 30 mins to 144 hr post treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on scale
Groups:
- Indomethacin Patch: Indomethacin patch to be applied on the sprained ankle BID
Arm/Group | Indomethacin Patch | Placebo Patch
Number analyzed (Participants) | 135 | 135
Score on scale
  0.5 hr | 6.90 (1.558) | 6.89 (1.329)
  1 hr | 6.85 (1.510) | 6.86 (1.407)
  2 hr | 6.55 (1.505) | 6.63 (1.485)
  4 hr | 6.26 (1.547) | 6.44 (1.609)
  8 hr | 6.30 (1.501) | 6.37 (1.667)
  12 hr | 5.88 (1.619) | 6.18 (1.757)
  24 hr | 5.27 (1.743) | 5.47 (1.876)
  36 hr | 4.62 (1.875) | 5.12 (1.933)
  48 hr | 4.40 (1.735) | 4.86 (1.805)
  60 hr | 4.08 (1.860) | 4.67 (1.886)
  72 hr | 3.76 (1.911) | 4.47 (1.825)
  84 hr | 3.48 (1.719) | 4.13 (1.804)
  96 hr | 3.21 (1.667) | 3.97 (1.902)
  108 hr | 3.22 (1.571) | 3.66 (1.843)
  120 hr | 2.95 (1.627) | 3.58 (1.814)
  132 hr | 2.84 (1.461) | 3.35 (1.804)
  144 hr | 2.70 (1.366) | 3.23 (1.713)

4. Secondary Outcome: Change From Baseline in NRS at Rest
Description: Mean changes in pain intensity at each time point at rest twice daily (in the morning and afternoon) from treatment day 1 to day 7 between treatment groups at time points 0.5 hrs, 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, 36 hrs, 48 hrs, 60 hrs, 72 hrs, 84 hrs, 96 hrs, 108 hrs, 120 hrs, 132 hrs and 144 hrs was measured using NRS. The NRS is a horizontal line with a scale from 0-10. After application of patch (indomethacin or reference patch), participants were asked to choose a number that relates to their pain intensity on the scale of 0 to 10, where 0 represents no pain and 10 represents the worst possible pain.
Time Frame: Baseline (Day 1) to Day 7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Indomethacin Patch | Placebo Patch
Number analyzed (Participants) | 135 | 135
Score on scale | -3.581 (0.1273) | -3.194 (0.1228)

5. Secondary Outcome: Time to Onset of Pain Relief
Description: Time to onset of pain relief was measured by the time to reach a pain relief score of "1" ("A little or perceptible pain relief").
Time Frame: Baseline (Day 1) to Day 3
Population: as for outcome 2
Measure: Median (Full Range); unit: Days
Arm/Group | Indomethacin Patch | Placebo Patch
Number analyzed (Participants) | 135 | 135
Days | 0.168 [0.09 to 0.19] | 0.208 [0.09 to 0.51]

6. Secondary Outcome: Assessment of Sum of Pain Intensity Difference (SPID) on Movement
Description: SPID was calculated as sum of products of Pain Intensity Differences (PID) at a given time-point (t) with the time-interval from that time-point to the previous time-point (t-1). The time-intervals used were 0 hrs (Day 1, pre treatment), 0.5 hrs, 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, 36 hrs, 48 hrs, 60 hrs, 72 hrs, 84 hrs, 96 hrs, 108 hrs, 120 hrs, 132 hrs and 144 hrs. Positive and higher scores indicate greater reduction in pain. SPIDt = ∑PID x (time t - time t-1).
  Pain Intensity was assessed at baseline and at each time-point based on numerical rating scale (NRS) which is a horizontal line with a scale from 0-10, where 0 represents "No" and 10 represents the "worst possible pain".
Time Frame: Baseline (Day 1) to Day 7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Indomethacin Patch | Placebo Patch
Number analyzed (Participants) | 135 | 135
Score on scale
  SPID (1-2 day) | 1.402 (0.0985) | 1.169 (0.0985)
  SPID (1-7 day) | 17.62 (0.7113) | 15.82 (0.7113)

7. Secondary Outcome: Sum of Pain Intensity Difference and Pain Relief (SPRID) on Movement
Description: SPRID:Sum of Pain Intensity Difference (SPID) and Total Pain Relief (TOTPAR) at each post-dosing time-point.
  SPRID score ranged from -5.8 (least pain relief) to 40.3 (highest pain relief). SPID and TOTPAR were calculated as weighted sums of Pain Intensity Differences (PID) and Pain Relief Scores (PRS) at each measurement time; 0 hr (Day 1, pre treatment), 0.5 hr, 1 hr, 2 hr, 4 hr, 8 hr, 12 hr, 24 hr, 36 hr, 48 hr, 60 hr, 72 hr, 84 hr, 96 hr, 108 hr, 120 hr, 132 hr and 144 hr, respectively.
  PID was derived by subtracting the pain severity score at a given post-dosing time-point from the baseline [based on NRS which is a horizontal line with a scale from 0-10. where 0 represents "No" and 10 represents the "worst possible pain"]. NR scores were converted into PID scores by subtracting them from baseline pain scores.
  PRS was assessed on 5-point categorical pain relief rating scale [0-no relief, 1-little relief, 2-some relief, 3-a lot of relief, 4-complete relief]
Time Frame: Baseline (Day 1) to Day 7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Indomethacin Patch | Placebo Patch
Number analyzed (Participants) | 135 | 135
Score on scale
  SPRID (1-2 days) | 2.594 (0.1608) | 2.099 (0.1608)
  SPRID (1-3 days) | 7.025 (0.3409) | 5.695 (0.3409)
  SPRID (1-7 days) | 28.85 (1.1045) | 25.43 (1.1045)

8. Secondary Outcome: Total Pain Relief (TOTPAR) on Movement
Description: TOTPAR was calculated as sum of products of pain relief (PR) at a given time-point (t) with the time-interval from that time-point to the previous time-point (t-1). The time-intervals used were 0 hrs (Day 1, baseline), 0.5 hrs, 1 hr, 2 hrs, 4 hrs, 8 hrs, 12 hrs, 24 hrs, 36 hrs, 48 hrs, 60 hrs, 72 hrs, 84 hrs, 96 hrs, 108 hrs, 120 hrs, 132 hrs and 144 hrs. Higher score indicated greater pain relief.
  TOTPARt = ∑PR x (time t - time t-1). PR score was assessed at each of the above time-points based on a 5-point categorical scale [0-no relief, 1-little relief, 2-meaningful relief, 3-a lot of relief, 4-complete relief].
Time Frame: Baseline (Day 1) to Day 7
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Score on scale
Arm/Group | Indomethacin Patch | Placebo Patch
Number analyzed (Participants) | 135 | 135
Score on scale
  TOPTAR (1-2 days) | 1.197 (0.0695) | 0.935 (0.0692)
  TOPTAR (1-3 days) | 3.057 (1.389) | 2.44 (0.1384)
  TOPTAR (1-7 days) | 11.27 (0.4234) | 9.649 (0.4218)

9. Secondary Outcome: Patients' Global Assessment to Treatment
Description: Patients global assessment in response to treatment was measured at the end of the study on a scale of 0 to 4 where: 0- Poor; 1- Fair; 2- Good; 3- Very Good; 4- Excellent
Time Frame: Baseline (Day 1) to Day 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Indomethacin Patch | Placebo Patch
Number analyzed (Participants) | 135 | 135
Score on scale | 2.7 (0.88) | 2.2 (0.08)

10. Secondary Outcome: Rate of Rescue Medication Use
Description: Rescue medication use was monitored throughout a period of 14 days.
Time Frame: Baseline (Day 1) to Day 14
Population: as for outcome 2
Measure: Number; unit: Number of participants
Arm/Group | Indomethacin Patch | Placebo Patch
Number analyzed (Participants) | 135 | 135
Number of participants | 4 | 7

11. Secondary Outcome: Time to First Dose of Rescue Medication Use
Description: Rescue medication use was monitored throughout a period of 14 days.
Time Frame: Baseline (Day 1) to Day 14
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Indomethacin Patch | Placebo Patch
Number analyzed (Participants) | 135 | 135
Days | 0.198 [0.06 to 0.25] | 0.681 [0.21 to 2.07]

12. Secondary Outcome: Total Dose of Rescue Medication Use
Description: Rescue medication use was monitored throughout a period of 14 days.
Time Frame: Baseline (Day 1) to Day 14
Population: as for outcome 2
Measure: Median (Full Range); unit: Dose
Arm/Group | Indomethacin Patch | Placebo Patch
Number analyzed (Participants) | 135 | 135
Dose | 3 [1 to 4] | 4 [1 to 10]

ADVERSE EVENTS:
Time Frame: 19 days
Arm/Group | Indomethacin Patch | Placebo Patch
Serious Adverse Events (participants affected / at risk) | 0/135 | 0/135
Other Adverse Events (participants affected / at risk) | 10/135 | 5/135
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Indomethacin Patch (N=135) | Placebo Patch (N=135)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Application site pruritis (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0)
Upper respiratory tract infections (Infections and infestations) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vascular rupture (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.